CLINICAL TRIAL: NCT03727230
Title: Single-arm Multicenter Clinical Trial of Blood Transfusion From RhD+ Donors to Asian-type DEL Recipients
Brief Title: RhD+ Blood Transfusion to Asian-type DEL Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Collaborators: Sun Yat-sen University (Other); Southern Medical University, China (Other); Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Guangdong Second Provincial General Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial Institute of Biological Products And Materia Medica (Other); Shenzhen Second People's Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEL
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-03

CONDITIONS: Blood Transfusion; Rhesus Isoimmunisation Due to Anti-D; Blood Group Antigen Abnormality
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Intervention Model Description: A single-arm clinical trial of Chinese Asian-type DEL patients receiving RhD+ RBC transfusion was conducted.
  Although truly RhD-negative patients receiving RhD+ RBC transfusion were recognized as the ideal control group, they were not included in this study because it did not comply with the Chinese Clinical Blood Transfusion Standard and ethics principles. The truly RhD-negative patients could receive RhD+ blood only in emergency situations under conditions of an insufficient stock of RhD-negative RBCs. Thus, the summarized alloanti-D rate (203/720, 28.2%; 95% CI, 19%-32%) in truly RhD-negative patients with similar mixed diseases after RhD+ RBC transfusion reported in the meta-analysis （Vox Sang 2021, http://doi.org/10.1111/vox.13232）was used as the control for comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asian-type DEL recipients (Experimental): First, to identify Asian-type DEL patients by phenotyping and genotyping methods in the Chinese recipients having a serologically apparent RhD-negative phenotype.
  Then, blood transfusion of RhD+ blood rather than rare RhD-negative blood to the Asian-type DEL recipients which met the inclusion criteria.
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Transfusion with RhD+ blood product rather than rare RhD-negative blood to Asian-type DEL recipients

SUMMARY:
Red blood cells (RBCs) from Asian-type DEL blood group express very weak RhD antigen and are falsely typed as RhD-negative blood group in routine RhD testing. Until now, Asian-type DEL (D-eluate) patients still be treated as rare RhD-negative patients in the clinic. Previous study from the Asian-type DEL pregnant women with RhD+ fetus showed no occurrence of alloanti-D immunization. This result, however, does not directly be applied for Asian-type DEL patients receiving RhD+ blood transfusions, as lacking of direct evidence regarding the safety and underlying mechanism.

In this study, the patients with Asian-type DEL were identified and received RhD+ blood transfusion, then evaluations of any adverse reactions, especially the active follow-up alloantibody test, were prospectively conducted.

DETAILED DESCRIPTION:
Red blood cells (RBCs) from Asian-type DEL individuals express very weak RhD antigen and are falsely typed as RhD-negative in routine RhD testing. Recent studies have shown that 9-30% of individuals with a serologically apparent RhD-negative phenotype in East and Southeast Asian populations, including Chinese, Korean, Japanese, Thai and Myanmar, actually are not truly RhD-negative but exhibit the DEL (D-eluate) phenotype, which represents almost 1.7 million Asian-type DEL individuals in China, 250,000 in Korea, Japan, Thailand, and Myanmar as well as at least 90,000 in the US among Asian immigrants. Nowadays, Asian-type DEL patients are conventionally transfused with RhD-negative RBC, which are difficult to organize because of the undersupply of the rare RhD-negative blood in these Asian countries, due to low frequency distribution (0.3-0.4%).

However, our previous study demonstrated that Asian-type DEL pregnant women with RhD+ fetus did not develop alloanti-D during the pregnancy. Latter, this phenomenon was confirmed by different medical centers in China. Accordingly, Asian-type DEL patients may also not be able to produce alloanti-D after transfusion with RhD+ RBC and consequently the use of RhD-negative RBCs for the transfusion management of Asian-type patients may be superfluous. However, this hypothesis needs to be carefully proved.

In this study, we were able to verify this assumption. Blood samples from 2,011 Chinese patients with a primary RhD-negative phenotype from the hospitals in Guangzhou of China were typed for Asian-type DEL blood group in the Guangzhou Blood Center. DEL phenotyping was performed by the serological adsorption/elution antibody testing and genotyping for the Asian-type DEL specific allele (RHD*1227A) detection was conducted using a well validated high-resolution melting (HRM) approach. Then, transfusions of RhD+ RBC were performed in a cohort of Asian-type DEL patients. After RhD+ blood transfusion, evaluations of any adverse reactions, especially the active follow-up alloantibody test, were conducted to evaluate the alloanti-D immunization. Besides, effectiveness of transfusion (Hb changes) was also recorded.

ELIGIBILITY:
Inclusion criteria for eligible participants were as follows: (1) Asian-type DEL blood group; (2) male patients, or female patients ≥ 49 years of age, or female with severe illness and no plan for further pregnancy; (3) needing blood transfusion in line with guidelines for internal medicine or surgery; and (4) signed voluntary informed consent for blood transfusion treatment before the trial.

The exclusion criteria were: (1) adverse reaction in a previous transfusion; (2) allergies to blood products or immunodeficiency diseases; (3) needing massive blood transfusion for acute blood loss; (4) positive pregnancy test results; (5) conscious dysfunction or severe mental illness; and (6) unsuitability for the study, as estimated by the principal investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligible participant inclusions were as follows: (1) all male Asian-type DEL patients; (2) female Asian-type DEL patients beyond the gestational age (≥49 years); (3) female Asian-type DEL patients of childbearing age but with severe illness and no plan of further pregnancy
Enrollment: 54 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongshui Fu, MD, PhD, Study Chair — Guangzhou Blood Center
Locations (10):
- China (10):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Blood Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Luo Y, Wen J, Sun Y, Jia S, Ou C, Yang W, Chen J, Ye H, Liu X, Liang Y, Lu Z, Feng Y, Wu X, Xiao M, Mo J, Zhou Z, Wang Z, Liao Z, Chen J, Wei L, Luo G, Santoso S, Fichou Y, Flegel WA, Shao C, Li C, Zhang R, Fu Y. Patients with Asian-type DEL can safely be transfused with RhD-positive blood. Blood. 2023 Apr 27;141(17):2141-2150. doi: 10.1182/blood.2022018152. PMID 36638337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ranged between October 2016 and November 2021 in all hospitals located in Guangzhou of China.
Pre-assignment Details: The enrolled participants are the Asian-type DEL patients with application for RBCs product from Guangzhou Blood Center, which is the only institute responsible for blood supply in Guangzhou city of China. Guangzhou is the capital city of Guangdong province in South China, with 15 million inhabitants.
  When any enrolled participants did not receive any blood transfusion finally, because of no need of blood transfusion in the clinic, they were excluded from the study.
Groups:
- Asian-type DEL Recipients: Asian-type DEL patients was identified by phenotyping and genotyping methods, then D+ RBCs rather than rare D-negative RBCs were transfused to the "Aisa type" DEL recipients.
Period: Overall Study
Arm/Group | Asian-type DEL Recipients
Started | 54
Completed | 42
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Groups:
- Asian-type DEL Recipients: After identification of Asian-type DEL patients by phenotyping and genotyping methods, then D+ RBCs rather than rare D-negative RBCs were transfused to the Aisa-type DEL recipients who met the inclusion criteria.
  Blood transfusion: Transfusion with D+ blood rather than the rare D-negative blood to Asian-type DEL recipients
Arm/Group | Asian-type DEL Recipients
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 54
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 54
Asian-type DEL patients received D+ RBC transfusion [Count of Participants; unit: Participants] | 54

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Alloanti-D Immunization in Asian-type DEL Recipients Transfused With RhD+ RBCs
Description: For the Chinese Asian-type DEL recipients identified by the serological adsorption/elution test and HRM genotyping analysis, RhD+ RBC transfusion was performed. Then, the new blood samples from the patients were obtained after transfusion of RhD+ RBCs. The clinical significant alloantibodies against the common antigens of RBC were re-tested by antibody screening test. And the antibody screening test was performed using ID-DiaCell I-II-III Asia Kit (BIO-RAD, Cressier, Switzerland) in saline by the tube method and an indirect antiglobulin test (IAT) with the DG Gel Coombs card (Diagnostic Grifols, Barcelona, Spain). Meanwhile, RhCE and Asian- type DEL typing were also tested again.
Time Frame: A median follow-up of 226 days (range, 32 to 1354 days) after RhD+ RBC transfusion
Measure: Count of Participants; unit: Participants
Groups:
- Asian-type DEL Recipients: After identification of Asian-type DEL patients by phenotyping and genotyping methods, then D+ RBCs rather than rare D-negative RBCs were transfused to the Aisan-type DEL recipients.
  Blood transfusion: Transfusion with D+ blood rather than the rare D-negative blood to Asian-type DEL recipients
Arm/Group | Asian-type DEL Recipients
Number analyzed (Participants) | 54
Participants
  No occurrence of alloanti-D immunization | 42
  Lost of follow-up | 12
Statistical Analysis 1: Comparison: Asian-type DEL Recipients; In this study, a single-arm clinical trial was conducted. The summarized alloanti-D rate (203/720, 28.2%; 95% CI, 19%-32%) in truly RhD-negative patients with similar mixed diseases after RhD+ RBC transfusion reported in the meta-analysis (Ji YL, et al. Vox Sang 2022; 117: 633-40) was used as the control for comparison with alloanti-D rate identified in Asian-type DEL patients after RhD+ RBC transfusion in the clinical trial; Test type: Other; p < 0.001, Chi-squared

2. Secondary Outcome: Adverse Transfusion Reaction Analysis in Asian-type DEL Recipients During or After RhD+ Blood Transfusion
Description: Matched D+ RBCs were provided to the 54 eligible Asian-type DEL patients by the Guangzhou Blood Center and transfused at their respective hospitals. Patients were monitored for any adverse events during transfusion and a few days thereafter, which mainly involved acute nor delayed hemolytic transfusion reactions, as well as nonhemolytic reactions, including allergic and febrile nonhemolytic reactions and circulatory overload during or after transfusion. If the symptoms of hemolysis were suspected, the laboratory biochemical measurements were also performed.
Time Frame: During the blood transfusion and in the days of hospitalization
Measure: Count of Participants; unit: Participants
Groups:
- Asian-type DEL Recipients: To identify Asian-type DEL patients by phenotyping and genotyping methods in the Chinese recipients and then blood transfusion of D+ blood rather than the rare D negative blood to the identified Aisan-type DEL recipients.
  Blood transfusion: Transfusion with D+ blood rather than the rare D negative blood to Asian-type DEL recipients
Arm/Group | Asian-type DEL Recipients
Number analyzed (Participants) | 54
Participants
  Without adverse transfusion reaction | 54
  With adverse transfusion reaction | 0

ADVERSE EVENTS:
Time Frame: Assessed up to 1354 days following transfusion, a median of 226 days
Description: In the condition of correct blood group typing and cross-matching before transfusion, and carefully checking and monitoring during the transfusion, the transfusion treatment is quite safe with very low frequency of serious adverse event and mortality.
Groups:
- Asian-type DEL Recipients: To identify Asian-type DEL patients by phenotyping and genotyping methods in the Chinese recipients and then blood transfusion of RhD+ blood rather than rare RhD-negative blood to the Aisan-type DEL recipients who met the inclusion criteria.
  Blood transfusion: Transfusion with RhD+ blood rather than rare RhD-negative blood to Asian-type DEL recipients
Arm/Group | Asian-type DEL Recipients
All-Cause Mortality (participants affected / at risk) | 7/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asian-type DEL Recipients (N=54)
Adverse blood transfusion reactions (General disorders) | 0 — Adverse blood transfusion reactions mainly include acute nor delayed hemolytic transfusion reactions, as well as nonhemolytic reactions, including allergic and febrile nonhemolytic reactions and circulatory overload during or after transfusion.

LIMITATIONS AND CAVEATS:
A large-scale clinical trial cannot be conducted since Asian-type DEL is rarely distributed in our population, with a frequency of approximately 0.1%. Additionally, a prudent inclusion criterion was adopted in this study to avoid potential alloanti-D immunization and negative influences on pregnancy in women of reproductive age and young girls, in which they were excluded from the trial with great caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03727230/Prot_SAP_000.pdf